CLINICAL TRIAL: NCT03681184
Title: ILLUMINATE-A: A Phase 3 Randomized, Double-Blind, Placebo-Controlled Study With an Extended Dosing Period to Evaluate the Efficacy and Safety of Lumasiran in Children and Adults With Primary Hyperoxaluria Type 1
Brief Title: A Study to Evaluate Lumasiran in Children and Adults With Primary Hyperoxaluria Type 1
Acronym: ILLUMINATE-A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALN-GO1-003; 2018-001981-40 (EudraCT Number)
Expanded Access: NCT04125472 (Approved for marketing)
Record Dates: First submitted 2018-09-19; First posted 2018-09-21 (Actual); Results first posted 2021-01-19 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-07

CONDITIONS: Primary Hyperoxaluria Type 1 (PH1)
Keywords: PH1; Primary hyperoxaluria; RNAi therapeutic; siRNA; AGT; Oxalate
MeSH Terms: conditions — Primary hyperoxaluria type 1; Hyperoxaluria, Primary | interventions — lumasiran

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo/Lumasiran (Placebo Comparator): Lumasiran-matching placebo (normal saline [0.9% NaCl]) was administered subcutaneously (SC) at Day 1 and Months 1, 2 and 3 during the 6-Month Double-blind (DB) Period, followed by lumasiran SC, 3.0 mg/kg, at Months 6, 7 and 8 during the 3-Month Blinded Treatment Extension Period, followed by lumasiran SC, 3.0 mg/kg, at Month 9 and then every three months during the 51-Month Open-label Extension (OLE) period.
  Interventions: Drug: Placebo; Drug: Lumasiran
- Lumasiran/Lumasiran (Experimental): Lumasiran was administered SC, 3.0 mg/kg, at Day 1 and Months 1, 2 and 3 during the 6-Month DB Period, followed by lumasiran SC, 3.0 mg/kg at Month 6, and lumasiran-matching placebo SC at Months 7 and 8 during the 3-Month Blinded Treatment Extension Period, followed by lumasiran SC, 3.0 mg/kg, at Month 9 and then every three months during the 51-Month OLE period.
  Interventions: Drug: Placebo; Drug: Lumasiran

INTERVENTIONS:
Drug: Placebo — Placebo by SC injection
Drug: Lumasiran — Lumasiran by SC injection
  Other Names: ALN-GO1

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of lumasiran in children and adults with primary hyperoxaluria type 1 (PH1).

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide written informed consent or assent and to comply with study requirements
* Confirmation of PH1 disease
* Meet the 24 hour urine oxalate excretion requirements
* If taking Vitamin B6 (pyridoxine), must have been on stable regimen for at least 90 days

Exclusion Criteria:

* Clinically significant health concerns (with the exception of PH1) or clinical evidence of extrarenal systemic oxalosis
* Clinically significant abnormal laboratory results
* Known active or evidence of HIV or hepatitis B or C infection
* An estimated GFR of < 30 mL/min/1.73m^2 at screening
* Received an investigational agent within 30 days or 5 half-lives before the first dose of study drug or are in follow-up of another clinical study
* History of kidney or liver transplant
* Known history of multiple drug allergies or allergic reaction to an oligonucleotide or GalNAc
* History of intolerance to subcutaneous injection
* Women who are pregnant, planning a pregnancy, or breast-feeding or those of child bearing potential and not willing to use contraception
* History of alcohol abuse within the last 12 months, or unable or unwilling to limit alcohol consumption throughout the study

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2024-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (16):
- United States (5):
  - Clinical Trial Site, San Diego, California
  - Clinical Trial Site, Jacksonville, Florida
  - Clinical Trial Site, Rochester, Minnesota
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Cleveland, Ohio
- France (2):
  - Clinical Trial Site, Lyon
  - Clinical Trial Site, Paris
- Clinical Trial Site, Bonn, Germany
- Israel (3):
  - Clinical Trial Site, Haifa
  - Clinical Trial Site, Jerusalem
  - Clinical Trial Site, Nahariya
- Clinical Trial Site, Amsterdam, Netherlands
- Clinical Trial Site, Bern, Switzerland
- Clinical Trial Site, Dubai, United Arab Emirates
- United Kingdom (2):
  - Clinical Trial Site, Birmingham
  - Clinical Trial Site, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Frishberg Y, Saland JM, Lieske JC, Du W, Coenen M, Hogan J, Sellier-Leclerc AL, Groothoff JW, Kaspar C, Gansner JM, Hulton SA; ILLUMINATE-A study investigators. Final Results of the ILLUMINATE-A Phase 3 Clinical Trial of Lumasiran for Primary Hyperoxaluria 1. Clin J Am Soc Nephrol. 2025 Dec 4. doi: 10.2215/CJN.0000000916. Online ahead of print. No abstract available. PMID 41343248
- [Derived] Garrelfs SF, Frishberg Y, Hulton SA, Koren MJ, O'Riordan WD, Cochat P, Deschenes G, Shasha-Lavsky H, Saland JM, Van't Hoff WG, Fuster DG, Magen D, Moochhala SH, Schalk G, Simkova E, Groothoff JW, Sas DJ, Meliambro KA, Lu J, Sweetser MT, Garg PP, Vaishnaw AK, Gansner JM, McGregor TL, Lieske JC; ILLUMINATE-A Collaborators. Lumasiran, an RNAi Therapeutic for Primary Hyperoxaluria Type 1. N Engl J Med. 2021 Apr 1;384(13):1216-1226. doi: 10.1056/NEJMoa2021712. PMID 33789010

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with PH1 were enrolled at sixteen sites in France, Germany, Israel, the Netherlands, Switzerland, the United Arab Emirates, the United Kingdom and the United States.
Pre-assignment Details: Participants were treated with placebo or lumasiran during the 6-month Double-Blind (DB) Period. All participants received lumasiran during the 3-Month Blinded Treatment Extension Period and 51-Month Open-Label Extension Period.
Period: 6-Month Double-Blind Period
Arm/Group | Placebo/Lumasiran | Lumasiran/Lumasiran
Started | 13 | 26
Completed | 13 | 25
Not Completed | 0 | 1
Not completed — Parent/Caregiver Withdrew Consent | 0 | 1
Period: 3-Month Blinded Extension Period
Arm/Group | Placebo/Lumasiran | Lumasiran/Lumasiran
Started | 13 | 24 (1 participant discontinued study drug and entered safety follow up after the DB period.)
Completed | 13 | 24
Not Completed | 0 | 0
Period: Open-Label Extension Period
Arm/Group | Placebo/Lumasiran | Lumasiran/Lumasiran
Started | 13 | 24
Completed | 13 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All randomized participants who received any amount of study drug, was used for all baseline characteristics, except for 24-hour urinary oxalate excretion corrected for body surface area (BSA), which used the Safety Analysis Set (SAS): All participants who received any amount of study drug.
Groups:
- Placebo/Lumasiran: Lumasiran-matching placebo was administered SC at Day 1 and Months 1, 2 and 3 during the 6-Month DB Period, followed by lumasiran SC, 3.0 mg/kg, at Months 6, 7 and 8 during the 3-Month Blinded Treatment Extension Period, followed by lumasiran SC, 3.0 mg/kg, at Month 9 and then every three months during the 51-Month OLE period.
- Total: Total of all reporting groups
Arm/Group | Placebo/Lumasiran | Lumasiran/Lumasiran | Total
Number analyzed (Participants) | 13 | 26 | 39
Age, Customized [Count of Participants; unit: Participants]
  6 to <12 Years | 7 | 9 | 16
  12 to <18 Years | 1 | 5 | 6
  18 to <65 Years | 5 | 12 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 8 | 18 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 3 | 6
  White | 9 | 21 | 30
  Other | 0 | 2 | 2
  More than one race | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 13 | 25 | 38
Age at Informed Consent [Mean (Standard Deviation); unit: years] | 17.0 (15.19) | 18.7 (11.52) | 18.1 (12.68)
24-Hour Urinary Oxalate Excretion Corrected for BSA [Mean (Standard Deviation); unit: mmol/24hr/1.73m^2] | 1.79 (0.68) | 1.83 (0.60) | 1.82 (0.62)
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 78.834 (29.9841) | 82.967 (25.5499) | 81.589 (26.7820)
24-hour Urinary Oxalate:Creatinine Ratio [Mean (Standard Deviation); unit: mmol/mmol] | 0.231 (0.1306) | 0.209 (0.1012) | 0.216 (0.1106)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in 24-hour Urinary Oxalate Excretion Corrected for Body Surface Area (BSA) From Baseline to Month 6
Description: Percent change in 24-hour urinary oxalate excretion corrected for BSA was estimated by an average percent change from baseline across Months 3 through 6. Only valid urine samples without any non-protocol-related issues were included in the analysis. A negative change from Baseline indicates a favorable outcome.
Time Frame: Baseline to Month 6
Population: FAS: All randomized participants who received any amount of study drug.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo/Lumasiran | Lumasiran/Lumasiran
Number analyzed (Participants) | 13 | 26
percent change | -11.8 (3.8) | -65.4 (2.9)
Statistical Analysis 1: Comparison: Placebo/Lumasiran vs Lumasiran/Lumasiran; The Mixed-Effect Model Repeated Measures (MMRM) includes fixed effects of treatment arms (lumasiran vs. placebo) and scheduled visits (months 3, 4, 5, and 6), baseline 24-hour urinary oxalate corrected for BSA as a continuous fixed covariate, and patient as a random effect. The variance-covariance matrix is assumed to be unstructured. Satterthwaite approximation is used to estimate denominator degrees of freedom; Test type: Superiority; p < 0.0001, MMRM — P=1.685E-14; Difference in Least Squares (LS) Mean = -53.546, 95% CI 2-sided [-62.314 to -44.778], Standard Error of Mean 4.3224

2. Secondary Outcome: Absolute Change in 24-hour Urinary Oxalate Corrected for BSA From Baseline to Month 6
Description: Absolute change in 24-hour urinary oxalate excretion corrected for BSA was estimated by an average absolute change from baseline across Months 3 through 6. Only valid urine samples without any non-protocol-related issues were included in the analysis. A negative change from Baseline indicates a favorable outcome.
Time Frame: Baseline to Month 6
Population: FAS: All randomized participants who received any amount of study drug.
Measure: Least Squares Mean (Standard Error); unit: mmol/24hr/1.73m^2
Arm/Group | Placebo/Lumasiran | Lumasiran/Lumasiran
Number analyzed (Participants) | 13 | 26
mmol/24hr/1.73m^2 | -0.27 (0.08) | -1.24 (0.06)
Statistical Analysis 1: Comparison: Placebo/Lumasiran vs Lumasiran/Lumasiran; The MMRM includes fixed effects of treatment arms (lumasiran vs. placebo) and scheduled visits (months 3, 4, 5, and 6), baseline 24-hour urinary oxalate corrected for BSA as a continuous fixed covariate, and patient as a random effect. The variance-covariance matrix is assumed to be unstructured. Satterthwaite approximation is used to estimate denominator degrees of freedom; Test type: Superiority; p < 0.0001, MMRM — P=1.225E-11; Difference in LS Mean = -0.975, 95% CI 2-sided [-1.177 to -0.772], Standard Error of Mean 0.0998

3. Secondary Outcome: Percent Change in 24-hour Urinary Oxalate:Creatinine Ratio From Baseline to Month 6
Description: Percent change in 24-hour urinary oxalate:creatine ratio was estimated by an average percent change from baseline across Months 3 through 6. A negative change from Baseline indicates a favorable outcome.
Time Frame: Baseline to Month 6
Population: FAS: All randomized participants who received any amount of study drug.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo/Lumasiran | Lumasiran/Lumasiran
Number analyzed (Participants) | 13 | 26
percent change | -10.8 (5.4) | -62.5 (4.0)
Statistical Analysis 1: Comparison: Placebo/Lumasiran vs Lumasiran/Lumasiran; The MMRM includes fixed effects of treatment arms (lumasiran vs. placebo) and scheduled visits (months 3, 4, 5, and 6), baseline 24-hour urinary oxalate:creatinine ratio as a continuous fixed covariate, and patient as a random effect. The variance-covariance matrix is assumed to be unstructured. Satterthwaite approximation is used to estimate denominator degrees of freedom; Test type: Superiority; p < 0.0001, MMRM — P=5.032E-10; Difference in LS Mean = -51.7718, 95% CI 2-sided [-64.2653 to -39.2784], Standard Error of Mean 6.16118

4. Secondary Outcome: Percentage of Participants With 24-hour Urinary Oxalate Level Corrected for BSA at or Below 1.5 x ULN at Month 6
Description: The upper limit of normal (ULN) = 0.514 mmol/24hr/1.73m^2 for 24-hour urinary oxalate excretion corrected for BSA.
Time Frame: Month 6
Population: Participants from the FAS (all randomized participants who received any amount of study drug) for whom data are available.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/Lumasiran | Lumasiran/Lumasiran
Number analyzed (Participants) | 13 | 25
percentage of participants | 0 | 84.0
Statistical Analysis 1: Comparison: Placebo/Lumasiran vs Lumasiran/Lumasiran; The proportion of participants (lumasiran vs. placebo) with 24-hour urinary oxalate ≤1.5 x ULN at Month 6 is analyzed using the Cochran-Mantel-Haenszel test, stratified by baseline 24-hour urinary oxalate corrected for BSA (≤1.70 mmol/24hr/1.73m^2 vs. >1.70 mmol/24hr/1.73m^2). The difference in proportion (lumasiran vs. placebo) and the corresponding 95% confidence interval are calculated using the Newcombe method, based on the Wilson score; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P=8.341E-07; Difference in Proportions = 0.84, 95% CI 2-sided [0.55 to 0.94]

5. Secondary Outcome: Percentage of Participants With 24-hour Urinary Oxalate Level Corrected for BSA at or Below ULN at Month 6
Description: The upper limit of normal (ULN) = 0.514 mmol/24hr/1.73m^2 for 24-hour urinary oxalate excretion corrected for BSA.
Time Frame: Month 6
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo/Lumasiran | Lumasiran/Lumasiran
Number analyzed (Participants) | 13 | 25
percentage of participants | 0 | 52.0
Statistical Analysis 1: Comparison: Placebo/Lumasiran vs Lumasiran/Lumasiran; The proportion of participants (lumasiran vs. placebo) with 24-hour urinary oxalate ≤ULN at Month 6 is analyzed using the Cochran-Mantel-Haenszel test, stratified by baseline 24-hour urinary oxalate corrected for BSA (≤1.70 mmol/24hr/1.73m^2 vs. >1.70 mmol/24hr/1.73m^2). The difference in proportion (lumasiran vs. placebo) and the corresponding 95% confidence interval are calculated using the Newcombe method, based on the Wilson score; Test type: Superiority; p = 0.0010, Cochran-Mantel-Haenszel; Difference in Proportions = 0.52, 95% CI 2-sided [0.23 to 0.70]

6. Secondary Outcome: Percentage Change in Plasma Oxalate From Baseline to Month 6
Description: Percent change in plasma oxalate (umol/L) was estimated by an average percent change from baseline across Months 3 through 6. A negative change from Baseline indicates a favorable outcome.
Time Frame: Baseline to Month 6
Population: Plasma Oxalate Analysis Set: all participants who received any amount of study drug and had baseline plasma oxalate level ≥1.5×lower limit of quantitation (LLOQ). LLOQ is 5.55 μmol/L.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo/Lumasiran | Lumasiran/Lumasiran
Number analyzed (Participants) | 10 | 23
percent change | -0.3 (4.3) | -39.8 (2.9)
Statistical Analysis 1: Comparison: Placebo/Lumasiran vs Lumasiran/Lumasiran; The MMRM includes fixed effects of treatment arms (lumasiran vs. placebo) and scheduled visits (months 3, 4, 5, and 6), baseline plasma oxalate as a continuous fixed covariate, and patient as a random effect. The variance-covariance matrix is assumed to be unstructured. Satterthwaite approximation is used to estimate denominator degrees of freedom; Test type: Superiority; p < 0.0001, MMRM — P=2.862E-08; Difference in LS Mean = -39.48, 95% CI 2-sided [-50.10 to -28.87], Standard Error of Mean 5.181

7. Secondary Outcome: Absolute Change in Plasma Oxalate From Baseline to Month 6
Description: Absolute change in plasma oxalate (umol/L) was estimated by an average percent change from baseline across Months 3 through 6. A negative change from Baseline indicates a favorable outcome.
Time Frame: Baseline to Month 6
Population: Plasma Oxalate Analysis Set: all participants who received any amount of study drug and had baseline plasma oxalate level ≥1.5×LLOQ. LLOQ is 5.55 μmol/L.
Measure: Least Squares Mean (Standard Error); unit: μmol/L
Arm/Group | Placebo/Lumasiran | Lumasiran/Lumasiran
Number analyzed (Participants) | 10 | 23
μmol/L | 1.3 (1.1) | -7.5 (0.8)
Statistical Analysis 1: Comparison: Placebo/Lumasiran vs Lumasiran/Lumasiran; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < 0.0001, MMRM — P=3.893E-07; Difference in LS Mean = -8.71, 95% CI 2-sided [-11.45 to -5.98], Standard Error of Mean 1.338

8. Secondary Outcome: Change in Estimated Glomerular Filtration Rate (eGFR) From Baseline to Week 2 and Months 1, 2, 3, 4, 5 and 6
Description: eGFR is calculated from serum creatinine based on the Modification of Diet in Renal Disease formula for patients ≥18 years of age and the Schwartz Bedside Formula for patients >1 year to <18 years of age at screening. Change from baseline to Month 6 is reported.
Time Frame: Baseline, Week 2, Months 1, 2, 3, 4, 5 and 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Placebo/Lumasiran | Lumasiran/Lumasiran
Number analyzed (Participants) | 13 | 25
mL/min/1.73m^2
  Week 2: number analyzed (Participants) | 13 | 24
  Week 2 | -5 (9) | -4 (9)
  Month 1: number analyzed (Participants) | 12 | 25
  Month 1 | -6 (7) | -2 (12)
  Month 2 | -5 (8) | -2 (15)
  Month 3 | -3 (6) | 0 (11)
  Month 4: number analyzed (Participants) | 12 | 25
  Month 4 | -4 (8) | -4 (10)
  Month 5 | -4 (7) | -6 (13)
  Month 6 | 0 (6) | -3 (11)

9. Secondary Outcome: Absolute Change in 24-hour Urinary Oxalate Excretion Corrected for BSA From Baseline in the Extension Period
Description: Absolute change in 24-hour urinary oxalate excretion corrected for BSA was estimated by an average absolute change from baseline in the extension periods. Only valid urine samples without any non-protocol-related issues were included in the analysis. A negative change from Baseline indicates a favorable outcome.
Time Frame: From Baseline to Month 54 and Month 60
Population: All Lumasiran Treated Set: All participants who received any amount of lumasiran including participants who took lumasiran during the 6-month double-blinded period and participants who initially took placebo during the 6-month double-blinded period and then switched to lumasiran during the extension period. Overall number analyzed is number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: mmol/24hr/1.73m^2
Arm/Group | Placebo/Lumasiran | Lumasiran/Lumasiran
Number analyzed (Participants) | 6 | 23
mmol/24hr/1.73m^2
  At Month 54 | -0.951 (0.6148) | -1.086 (0.7678)
  At Month 60: number analyzed (Participants) | 0 | 19
  At Month 60 |  | -1.129 (0.7581)

10. Secondary Outcome: Percentage Change in 24-hour Urinary Oxalate Excretion Corrected by BSA From Baseline in the Extension Period
Description: Percent change in 24-hour urinary oxalate excretion corrected for BSA was estimated by an average percent change from baseline in the extension periods. Only valid urine samples without any non-protocol-related issues were included in the analysis. A negative change from Baseline indicates a favorable outcome.
Time Frame: From Baseline to Month 54 and Month 60
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo/Lumasiran | Lumasiran/Lumasiran
Number analyzed (Participants) | 6 | 23
percent change
  At Month 54 | -55.57 (11.903) | -53.87 (41.919)
  At Month 60: number analyzed (Participants) | 0 | 19
  At Month 60 |  | -53.98 (28.476)

11. Secondary Outcome: Percentage of Time That 24-hour Urinary Oxalate is at or Below 1.5 × ULN During Lumasiran Treatment
Description: The upper limit of normal (ULN) = 0.514 mmol/24hr/1.73m^2 for 24-hour urinary oxalate excretion corrected for BSA.
Time Frame: Up to Month 60
Population: All Lumasiran Treated Set: All participants who received any amount of lumasiran including participants who took lumasiran during the 6-month double-blinded period and participants who initially took placebo during the 6-month double-blinded period and then switched to lumasiran during the extension period.
Measure: Median (Full Range); unit: percentage of time
Arm/Group | Placebo/Lumasiran | Lumasiran/Lumasiran
Number analyzed (Participants) | 13 | 26
percentage of time | 89.44 [21.1 to 99.3] | 89.23 [1.7 to 98.6]

12. Secondary Outcome: Absolute Change in 24-hour Urinary Oxalate:Creatinine Ratio From Baseline in the Extension Period
Description: Absolute change in 24-hour urinary oxalate:creatinine ratio was estimated by an average absolute change from baseline to the end of the OLE period at Month 54 and Month 60. A negative change from Baseline indicates a favorable outcome.
Time Frame: From Baseline to Month 54 and Month 60
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mmol/mmol
Arm/Group | Placebo/Lumasiran | Lumasiran/Lumasiran
Number analyzed (Participants) | 6 | 24
mmol/mmol
  At Month 54 | -0.145 (0.1242) | -0.127 (0.1063)
  At Month 60: number analyzed (Participants) | 0 | 19
  At Month 60 |  | -0.138 (0.1162)

13. Secondary Outcome: Change in Estimated Glomerular Filtration Rate (eGFR) From Baseline in the Extension Period
Description: eGFR is calculated from serum creatinine based on the Modification of Diet in Renal Disease formula for patients ≥18 years of age and the Schwartz Bedside Formula for patients >1 year to <18 years of age at screening.
Time Frame: From Baseline to Month 54 and Month 60
Population: All Lumasiran Treated Set: All participants who received any amount of lumasiran including participants who took lumasiran during the 6-month double-blinded period and participants who initially took placebo during the 6-month double-blinded period and then switched to lumasiran during the extension period. Overall number analyzed is number of participants with data available for analysis. Number analysed is the number of participants with data available for analysis at the specified timepoint.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Placebo/Lumasiran | Lumasiran/Lumasiran
Number analyzed (Participants) | 6 | 23
mL/min/1.73m^2
  At Month 54 | -12.860 (9.5386) | -6.899 (12.9302)
  At Month 60: number analyzed (Participants) | 0 | 18
  At Month 60 |  | -2.892 (11.6544)

14. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical investigational participant administered a medicinal product & which does not necessarily have a causal relationship with this treatment. SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires in-patient hospitalization/prolongation of existing hospitalization, results in persistent/significant disability or incapacity, is a congenital anomaly or birth defect, is an important medical event that may not be immediately life-threatening/result in death/hospitalization but may jeopardize the participant & may require intervention to prevent one of the other outcomes listed above. All Lumasiran Treated Set: All participants who received any amount of lumasiran including participants who took lumasiran during 6-month double-blinded period & participants who initially took placebo during the 6-month double-blinded period and then switched to lumasiran during the extension period.
Time Frame: DB Period (Placebo): From first dose of study drug (Day 1) up to Month 6; Placebo/Lumasiran: From first dose of lumasiran (Month 6) up to end of study (Month 60); Lumasiran/Lumasiran: From first dose of lumasiran (Day 1) up to end of study (Month 60).
Population: Per the SAP, long-term safety of lumasiran (in the extension period [EP]) was to be summarized by treatment sequence (placebo/lumasiran & lumasiran/lumasiran) using the All Lumasiran Treated Set. In this set, data is presented during lumasiran treatment only. The lumasiran/lumasiran arm received lumasiran in both DB & EP period hence, safety data is reported together for DB+EP period for this arm. Placebo/Lumasiran: first day of lumasiran dosing (Month 6) was considered baseline (Day 1) of EP.
Measure: Count of Participants; unit: Participants
Groups:
- DB Period: Placebo: Lumasiran-matching placebo was administered SC at Day 1 and Months 1, 2 and 3 during the 6-Month DB Period.
Arm/Group | DB Period: Placebo | Placebo/Lumasiran | Lumasiran/Lumasiran
Number analyzed (Participants) | 13 | 13 | 26
Participants
  Adverse Event (AE) | 9 | 12 | 25
  Serious Adverse Event (SAE) | 0 | 1 | 5

15. Other Pre Specified Outcome: Rate of Renal Stone Events
Description: A renal stone event is defined as a patient-reported event that includes ≥1 of the following: visit to healthcare provider because of a renal stone; medication for renal colic; stone passage; macroscopic hematuria due to a renal stone. Lower rates indicate a favorable outcome.
Time Frame: 12-Month Period prior to Informed Consent, 6-Month DB Period
Population: FAS: All randomized participants who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: events per person-year
Arm/Group | Placebo/Lumasiran | Lumasiran/Lumasiran
Number analyzed (Participants) | 13 | 26
events per person-year
  12-Month Period prior to Informed Consent | 0.54 [0.26 to 1.13] | 3.19 [2.57 to 3.96]
  6-Month DB Period | 0.66 [0.25 to 1.76] | 1.09 [0.63 to 1.87]

16. Other Pre Specified Outcome: Change From Baseline in Nephrocalcinosis as Assessed by Renal Ultrasound
Description: Renal ultrasound data were used to grade medullary nephrocalcinosis findings (range: 0 to 3), where a higher grade indicates greater severity. Improving=if both sides improve, or one side improves and the other side has no change; No change=if both sides have no change; Worsening=if both sides worsen, or one side worsens and the other side has no change; Indeterminate=if one side improves and the other side worsens.
Time Frame: Baseline, Month 6
Population: Participants from the FAS (all randomized participants who received any amount of study drug) with both Baseline and Month 6 renal ultrasounds.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/Lumasiran | Lumasiran/Lumasiran
Number analyzed (Participants) | 12 | 22
Participants
  Improving | 0 | 3
  No Change | 11 | 19
  Worsening | 1 | 0
  Indeterminate | 0 | 0

ADVERSE EVENTS:
Time Frame: DB Period (Placebo): From first dose of study drug (Day 1) up to Month 6; Placebo/Lumasiran: From first dose of lumasiran (Month 6) up to end of study (Month 60); Lumasiran/Lumasiran: From first dose of lumasiran (Day 1) up to end of study (Month 60).
Description: Per the SAP, long-term safety of lumasiran (in the extension period [EP]) was to be summarized by treatment sequence (placebo/lumasiran & lumasiran/lumasiran) using the All Lumasiran Treated Set. In this set, data is presented during lumasiran treatment only. The lumasiran/lumasiran arm received lumasiran in both DB & EP period hence, safety data is reported together for DB+EP period for this arm. Placebo/Lumasiran: first day of lumasiran dosing (Month 6) was considered baseline (Day 1) of EP.
Groups:
- Placebo: Lumasiran-matching placebo was administered SC at Day 1 and Months 1, 2 and 3 during the 6-Month DB Period.
Arm/Group | Placebo | Placebo/Lumasiran | Lumasiran/Lumasiran
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/13 | 5/26
Other Adverse Events (participants affected / at risk) | 9/13 | 12/13 | 25/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=13) | Placebo/Lumasiran (N=13) | Lumasiran/Lumasiran (N=26)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Post procedural infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
Follicular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=13) | Placebo/Lumasiran (N=13) | Lumasiran/Lumasiran (N=26)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 8
Injection site erythema (General disorders) | 0 | 1 | 3
Injection site reaction (General disorders) | 0 | 5 | 9
Otitis media acute (Infections and infestations) | 1 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2
Rhinitis (Infections and infestations) | 2 | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 3
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1 | 0
Thalassaemia beta (Congenital, familial and genetic disorders) | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1
Blepharitis (Eye disorders) | 0 | 0 | 1
Dacryostenosis acquired (Eye disorders) | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 2 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Gingival hypertrophy (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2 | 2
Asthenia (General disorders) | 0 | 0 | 1
Catheter site extravasation (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 2
Influenza like illness (General disorders) | 0 | 1 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 2 | 3
Vaccination site pain (General disorders) | 0 | 0 | 3
Vaccination site swelling (General disorders) | 0 | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1 | 1
Immunisation reaction (Immune system disorders) | 0 | 1 | 2
Milk allergy (Immune system disorders) | 0 | 0 | 1
Asymptomatic COVID-19 (Infections and infestations) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 4 | 4
Cellulitis (Infections and infestations) | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 1 | 1
Fungal foot infection (Infections and infestations) | 0 | 0 | 1
Fungal skin infection (Infections and infestations) | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 1 | 0
Herpes simplex reactivation (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Infected bite (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 4
Onychomycosis (Infections and infestations) | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1 | 0
Pyelitis (Infections and infestations) | 0 | 1 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1 | 1
Tooth infection (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 3
Viral infection (Infections and infestations) | 0 | 1 | 0
Viral sinusitis (Infections and infestations) | 0 | 0 | 1
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Nail injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 2
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Cardiac murmur (Investigations) | 0 | 0 | 1
Electrocardiogram ST segment depression (Investigations) | 0 | 1 | 0
Electrocardiogram T wave inversion (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Protein urine present (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 2 | 1
Weight gain poor (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 2
Headache (Nervous system disorders) | 3 | 2 | 5
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 1 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 1
Post abortion haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 1
Enuresis (Psychiatric disorders) | 0 | 0 | 1
Fear of injection (Psychiatric disorders) | 0 | 0 | 1
Irritability (Psychiatric disorders) | 0 | 0 | 1
Separation anxiety disorder (Psychiatric disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 3
Haematuria (Renal and urinary disorders) | 0 | 1 | 1
Hypertonic bladder (Renal and urinary disorders) | 0 | 0 | 1
Hypocitraturia (Renal and urinary disorders) | 0 | 1 | 0
Microalbuminuria (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 2
Polyuria (Renal and urinary disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Renal cyst (Renal and urinary disorders) | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1
Renal pain (Renal and urinary disorders) | 0 | 1 | 3
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Priapism (Reproductive system and breast disorders) | 0 | 1 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Actinic cheilitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 3
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Livedo reticularis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 1
White coat hypertension (Vascular disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 2
Injection site discomfort (General disorders) | 0 | 0 | 2
Injection site pain (General disorders) | 0 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-05-06): https://cdn.clinicaltrials.gov/large-docs/84/NCT03681184/Prot_002.pdf
  • Statistical Analysis Plan (2019-11-21): https://cdn.clinicaltrials.gov/large-docs/84/NCT03681184/SAP_001.pdf